CLINICAL TRIAL: NCT06043037
Title: Peri-implant Soft and Hard Tissue Changes Around Maxillary Anterior Immediate Implants Using Socket Shield Technique Versus a Combination of Socket Shield Technique and Autogenous Demineralized Dentin Graft: Randomized Clinical Trial
Brief Title: Elamrousy Modified Approach for Socket Shield Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Assistant Professor of periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-82
Record Dates: First submitted 2023-07-15; First posted 2023-09-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Implant Site Reaction; Tooth Extraction Status Nos; Dental Implant Failed

STUDY DESIGN:
Intervention Model Description: The present study included 50 participants, aged 20 to 45, with teeth that needed to be extracted. After Kafrelsheikh University research ethics committee approval, participants were randomized into 2 groups: the control group patients underwent immediate implantation using SS protocol, while the study group patients underwent the same procedure, but ADDG was created using the extracted palatal portion of the tooth; and then placed in the peri-implant gap defect. Clinically, pink aesthetic score (PES), midfacial mucosal alterations (MFMA), implant stability quotient (ISQ) were observed at baseline, six and twelve months after implantation. Moreover, baseline, 6- and 12-months alterations of radiographic horizontal bone dimension (HBD), buccal marginal bone level (BMBL), peri-implant Bone Density (PIBD) and peri-implant vertical bone defect (PIVBD) changes were assessed using cone beam computed tomography (CBCT).
Who Masked: Participant, Outcomes Assessor
Masking Description: neither participant nor the outcome assessor know the group districution
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Implant Placement Using Socket Shield Technique with autogenous demineralized dentin graft (Active Comparator): after immediate implantation using Socket Shield Technique, the palatal root portion will be converted to autogenous demineralized dentin graft and used for grafting the defect between the socket shield and the implant fixture
  Interventions: Procedure: Elamrousy Novel Approach for Immediate Implant Placement Using Socket Shield Technique
- Immediate Implant Placement Using Socket Shield Technique only without grafting the defect (Experimental): after insertion of immediate implant Using Socket Shield Technique, the bone defect between the socket shield and the implant fixture will be left ungrafted
  Interventions: Procedure: Immediate Implant Placement Using Socket Shield Technique alone

INTERVENTIONS:
Procedure: Elamrousy Novel Approach for Immediate Implant Placement Using Socket Shield Technique — The flapless strategy was used. To prepare the SS, tooth decoronation followed by root splitting mesio-distally. The palatally splitted portion of the root is atraumatically extracted while the intact buccal root portion is kept in place with thickness of 1.5mm.(12) The implant fixture is then placed palatally with 2mm gap distance in between. finally, that gap was grafted with ADDG
  Other Names: Immediate Implant Placement Using Socket Shield Technique grafted by autogenous demineralized dentin graft
  Arms: Immediate Implant Placement Using Socket Shield Technique with autogenous demineralized dentin graft
Procedure: Immediate Implant Placement Using Socket Shield Technique alone — The flapless strategy was used. To prepare the SS, tooth decoronation followed by root splitting mesio-distally. The palatally splitted portion of the root is atraumatically extracted while the intact buccal root portion is kept in place with thickness of 1.5mm.(12) The implant fixture is then placed palatally with 2mm gap distance in between. finally, that gap was left without grafts.
  Arms: Immediate Implant Placement Using Socket Shield Technique only without grafting the defect

SUMMARY:
The current trial aim was to evaluate clinically and radiographically the changes around dental implants inserted immediately in maxillary anterior esthetic zone using a novel combination of autogenous demineralized dentin graft (ADDG) with socket shield technique (SST) and compared this approach to socket shield technique (SST) alone.

The present study included 50 participants, aged 20 to 45, with teeth that needed to be extracted. After Kafrelsheikh University research ethics committee approval, participants were randomized into 2 groups: the control group patients underwent immediate implantation using SS protocol, while the study group patients underwent the same procedure, but ADDG was created using the extracted palatal portion of the tooth; and then placed in the peri-implant gap defect.

DETAILED DESCRIPTION:
However, Immediate placement protocol of dental implants reported favorable improvement of esthetic indices such as the Pink Esthetic Score (PES), mid-facial mucosal recession (MFMR) was the most common esthetic drawback. MFMR occurrences increase in case of thin gingival biotype, facial implant malposition, and thin or destroyed facial bone plate after tooth removal.

To avoid MFMR, dental implants should be placed immediately only when the clinical conditions are ideal including completely intact facial plate of bone, more than 1mm thick facial plate of bone, absence of periapical pathosis or infection at the extracted socket, thick gingival biotype, presence of sufficient bone palatal and apical to the extraction socket for proper positioning of the implant fixture and obtaining acceptable primary stability. These ideal conditions are rarely observed in the maxillary anterior region. Although proper patients' selection and treatment by specialists with high experience and skills, the esthetic outcomes of immediately placed dental implant showed unsatisfactory deteriorated facial tissues on the mid- to long-term.

Following root extraction, the thin delicate avascular cortical bone plate showed massive loss and deterioration due to loss of its vascular blood supply obtained from the root periodontal ligament. To overcome this negative esthetic outcome during immediate placement of dental implants, different materials and techniques were used around implants such as bone graft substitutes, growth factors and barrier membranes.

In 2010, Hurzeler and colleagues introduced a novel approach for immediate implantation called Socket Shield Technique (SST). This minimal invasive technique resulted in preservation of facial bone plate which in turn improved the esthetic outcomes. Partial extraction therapy, the root membrane technique and the modified SST are different terminologies and modifications of the original approch. In SST protocol, tooth decoronation followed by root splitting mesio-distally. The palatally splitted portion of the root is atraumatically extracted while the intact buccal root portion is kept in place with thickness of 1.5mm. The implant fixture is then placed palatally with 2mm gap distance in between. finally, that gap might be grafted or left without grafts.

SST showed enhancement of hard and soft tissue conditions around implants, implant stability and esthetic results compared with traditional immediate placement protocol of dental implants. Till now, few studies evaluated the effect of grafting the gap between the buccal tooth shield and the implant fixture.

Globally, extracted teeth are regarded as infectious waste. Teeth are made up of organic matrix and inorganic hydroxyapatite reinforcing phase, that's why teeth are gaining popularity as a potential resource for alveolar bone repair. Non-demineralized tooth grafts produced positive outcomes, but bone and tooth demineralization enhances the bioavailability of non-collagenous proteins associated with the matrix, such as osteocalcin, osteonectin, bone sialoprotein, phosphophoryn, and bone morphogenetic protein, which could promote the creation of new bone. A valuable three-dimensional biological scaffold with osteopromotive and osteoconductive properties is provided by ADDG. Additionally, it saves the patient money on the cost of other graft materials and lowers the worldwide amount of infectious dental waste.

The specific question of the current research was: Does using ADDG for grafting the gap between the tooth shield and the implant fixture in immediate dental implantation with SST improve the clinical and radiographic outcomes in comparison to immediate implant placement with SST alone without using bone graft?

ELIGIBILITY:
Inclusion Criteria:

* above the age of 18years
* presence of non-restorable maxillary anterior tooth
* had intact socket walls following tooth extraction
* the gingival biotype was thick.

Exclusion Criteria:

* history of systemic condition
* history of using bisphosphonates or other drugs that might impact bone turnover
* a history of smoking during the previous five years,
* a history of any acute infections at the surgical site,
* teeth having root resorptions
* massive periodontal destruction
* buccally fractured root either vertically or horizontally beneath the alveolar crest.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Implant Stability Quotient (ISQ) | 24-month.
  Osstell TM was used to record the primary stability.ISQ, or Implant Stability Quotient, is a scale from 1 to 100 and is a measure of the stability of an implant. The ISQ scale has a non-linear correlation to micro mobility. With more than 1400 scientific references, we now know that high stability means >70 ISQ, between 60-69 is medium stability and < 60 ISQ is considered as low stability.
PES | 24months
  The pink esthetic score (PES) evaluates the esthetic outcome of soft tissue around implant-supported single crowns in the anterior zone by awarding seven points for the mesial and distal papilla, soft-tissue level, soft-tissue contour, soft-tissue color, soft-tissue texture, and alveolar process deficiency.Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value, the maximum achievable PES was 14.
Midfacial Mucosal Alterations | 24months
  , digital intraoral scans were recorded. To quantify the vertical changes in the soft tissues around implants buccally, the collected scans were digitally superimposed via matching Gom inspect software

SECONDARY OUTCOMES:
buccal marginal bone level (BMBL) | 24 months
  Utilizing CBCT sagittal sections, the BMBL was evaluated by computerized analysis. Navigation was done on the multiplanar display until the implant's precise same-view location was established on the reformatted cross-sectional section and panoramic view.

CONTACTS AND LOCATIONS:
Overall Officials: Walid AH Elamrousy, PhD, Principal Investigator — Faculty of Oral and Dental Medicine, Kafrelsheikh University
Locations (1):
- oral medicine and periodontology outpatient clinic, faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No